CLINICAL TRIAL: NCT01556243
Title: Impact of Breast Conservation Surgery on Surgical Outcomes and Cosmesis in Patients With Multiple Ipsilateral Breast Cancers (MIBC)
Brief Title: Breast-Conserving Surgery and Radiation Therapy in Patients With Multiple Ipsilateral Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACOSOG-Z11102; ACOSOG-Z11102; CDR0000728605 (Registry Identifier: NCI Physician Data Query); NCI-2012-00707 (Registry Identifier: NCI Clinical Trial Reporting Program)
Record Dates: First submitted 2012-03-15; First posted 2012-03-16 (Estimated); Results first posted 2023-11-30 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Breast Cancer
Keywords: stage IA breast cancer; stage IB breast cancer; stage II breast cancer; ductal breast carcinoma in situ; lobular breast carcinoma in situ
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Intraductal, Noninfiltrating; Breast Carcinoma In Situ

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Breast conservation surgery and radiation therapy (Experimental): Patients undergo breast conserving surgery. Patients receive adjuvant chemotherapy at the physician's discretion. Patients receiving chemotherapy will start treatment within 12 weeks following surgery. Patients receive radiation therapy within 8 weeks following the last dose of chemotherapy or within 10 weeks following surgery if not receiving chemotherapy. Patients receive endocrine therapy at the physician's discretion. Patient observation will occur every 6 months until 5 years after the end of radiation therapy.
  Interventions: Procedure: therapeutic conventional surgery; Radiation: whole breast irradiation

INTERVENTIONS:
Procedure: therapeutic conventional surgery
Radiation: whole breast irradiation

SUMMARY:
RATIONALE: Breast-conserving surgery is a less invasive type of surgery for breast cancer and may have fewer side effects and improve recovery. Radiation therapy uses high-energy x rays to kill tumor cells. Giving radiation therapy after surgery may kill any tumor cells that remain after surgery.

PURPOSE: This phase II trial studies how well breast-conserving surgery and radiation therapy work in treating patients with multiple ipsilateral breast cancer

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To assess the local recurrence (LR) rate with breast-conservation in patients with multiple ipsilateral primary breast cancer (MIBC).

Secondary

* To examine the conversion rate to mastectomy secondary to persistent positive margins; poor cosmesis within the first year of attempting breast-conservation surgery (BCS) or inability to satisfy the radiation dose constraints on the boost to the lumpectomy bed of each site of disease.
* To assess whether patients who did not undergo re-excision for close margins (< 2 mm) have a higher local recurrence (LR) rate than patients for whom negative margins were achieved.
* To assess patient's perception of cosmesis and incidence of breast lymphedema.
* To assess incidence of breast lymphedema
* To examine the type and severity of adverse effects of breast conserving surgery and radiation for women with multiple ipsilateral primary breast cancer (MIBC).
* To examine the radiation-related side effects of whole-breast radiation with a boost to 1 large or > 1 lumpectomy site.

OUTLINE: This is a multicenter study.

Patients undergo breast-conserving surgery (BCS) with all lesions resected to negative margins using 1 lumpectomy or 2-3 separate lumpectomy incisions at the discretion of the surgeon. Patients receive adjuvant chemotherapy and/or endocrine therapy at the discretion of the treating medical oncologist based on tumor characteristics.

ELIGIBILITY:
Registration Inclusion Criteria:

1. Age ≥ 40 years per National Comprehensive Cancer Network (NCCN) recommendations for breast conservation.
2. Life Expectancy of at least 5 years, excluding diagnosis of breast cancer (Comorbid conditions should be taken into consideration, but breast cancer diagnosis is not a consideration)
3. Female Gender - Men are excluded from this study. Male breast cancer is a rare event.

   Men are rarely candidates for breast conservation surgery due to small breast size. Men are less likely to be candidates for breast conservation surgery if found to have MIBC.

   Men are rarely candidates for breast conservation surgery due to small breast size. Men are less likely to be candidates for breast conservation surgery if found to have MIBC.
4. Foci of Breast Cancer

   4.1 Upon clinical exam and pre-operative imaging by mammogram +/- MRI, two or three foci of biopsy proven breast cancer separated by > 2 cm of normal breast tissue.

   4.2 Foci must include at least one focus of invasive breast carcinoma with another focus of either invasive breast carcinoma or ductal carcinoma in situ (DCIS).

   No more than 2 quadrants with biopsy proven breast cancer.

   4.3 Note: The shortest distance between lesions must be reported on mammogram +/- MRI and eligibility criteria must be met on both, if both are obtained.

   4.4 Note: Patient is eligible for study if lesion is not visualized on all imaging modalities (i.e., any of the lesion(s) is/are visualized on MRI but not on mammogram OR visualized on mammogram but not on MRI).

   4.5 Ultrasound cannot be used to determine patient eligibility; eligibility to be determined by bilateral mammogram +/- MRI only.

   4.6 Fine needle aspirate of the second or third lesion to document malignancy is allowed if the first focus is shown to be invasive by core needle biopsy.

   4.7 Patient may remain on study if, upon pathological assessment, two or three lesions identified on pre-operative imaging represent one contiguous lesion.
5. Patients may be registered AFTER surgery and PRIOR TO radiation therapy if either of the criteria is met:

   5.1 An area of atypia > 2cm from the index lesion excised at the time of cancer operation is upgraded to DCIS or invasive carcinoma thereby identifying MIBC. OR

   5.2 Patient underwent resection of two or three foci of malignancy by breast conservation surgery with a minimum of one invasive focus of breast cancer and a minimum of 2 cm of normal breast tissue between the lesions on final pathology.
6. Mammogram Imaging - Bilateral mammogram ≤ 90 days prior to date of surgery.

   6.1 Note: For patients undergoing more than 1 breast operation, this is the date of the first breast surgery for breast cancer treatment.
7. Staging of Cancer - cN0 or cN1 disease
8. ECOG Performance Status (PS) - 0, 1, or 2.
9. Ability to Complete Questionnaires - Ability to complete questionnaire(s) by themselves or with assistance
10. Ability to Provide Written Informed Consent
11. Willing to Return to Enrolling Institution - Willing to return to enrolling institution for follow-up during the Active Monitoring Phase (the active treatment and observation portions) of the study. Patients are encouraged to return to the enrolling institution; however, patients may receive radiation therapy at a different institution other than the enrolling institution.

Registration Exclusion Criteria:

1. Pregnancy, Nursing and Requirement for Contraception - Pregnant women, nursing women and women of childbearing potential who are unwilling to employ adequate contraception (as determined by the treating physician) are excluded from participation.

   This study involves radiation therapy (WBI) that has known genotoxic, mutagenic and teratogenic effects.
2. Size of Single Focus of Disease on Preoperative Imaging - Largest single focus of disease > 5 centimeters by either mammogram or MRI or both. Note: Measurement of the largest single focus should include any satellite lesions within 1 centimeter of the index lesion.
3. Prior Staging Procedure - Surgical axillary staging procedure prior to first definitive breast operation. Note: FNA or core needle biopsy of axillary node is permitted.
4. Evidence of Metastatic Disease - Clinical or radiographic evidence of metastatic disease
5. Prior History of Breast Cancer - Prior history of ipsilateral breast cancer [DCIS, LCIS (lobular cancer in situ) or invasive]
6. Staging of Cancer - cNX, cN2, or cN3 disease
7. Breast Implants - Breast implants at time of diagnosis. Note: Patients who have had implants previously removed prior to diagnosis are eligible.
8. Systemic Illnesses or Concurrent Disease - Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would interfere significantly with whole breast irradiation (such as connective tissue disorders, lupus, scleroderma).
9. Uncontrolled Intercurrent Illness - Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
10. Bilateral Breast Cancer - Prior or current LCIS, DCIS or invasive breast cancer in the opposite breast (i.e., bilateral disease is not allowed).
11. Disallowed Prior Treatments - Treatment including radiation therapy, chemotherapy, biotherapy, hormonal therapy for this cancer prior to surgery (i.e., any neoadjuvant chemotherapy or endocrine therapy is not allowed). Patients who undergo surgical resection with breast conservation and then are treated with adjuvant systemic therapy are eligible to enroll prior to the start of radiotherapy.
12. Partial Breast Radiation - Planned partial breast radiation.
13. Known BRCA Mutations - Patients with known BRCA mutations. Patients who are not tested or whose testing result is not returned at the time of registration are not excluded from registering to this study.
14. Other Active Malignancies - Other active malignancy ≤ 5 years prior to registration.

14.1 Exceptions: Non-melanotic skin cancer or carcinoma-in-situ of the cervix.

14.2 Note: If there is a history of prior malignancy, they must not be receiving other specific treatment for their cancer.

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Actual)
Dates: Start 2012-07; Primary Completion 2022-06-01 (Actual); Study Completion 2023-04-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Judy Boughey, MD, Study Chair — Mayo Clinic
Locations (350):
- United States (350):
  - CHI Saint Vincent Cancer Center Hot Springs, Hot Springs, Arkansas
  - Epic Care-Dublin, Dublin, California
  - Bay Area Breast Surgeons, Incorporated, Emeryville, California
  - Epic Care Partners in Cancer Care, Emeryville, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Contra Costa Regional Medical Center, Martinez, California
  - Alta Bates Summit Medical Center-Summit Campus, Oakland, California
  - Bay Area Tumor Institute, Oakland, California
  - Stanford Cancer Institute, Palo Alto, California
  - Naval Medical Center-San Diego, San Diego, California
  - University of Colorado Cancer Center-Anschutz Cancer Pavilion, Aurora, Colorado
  - Catholic Health Initiatives NCORP, Englewood, Colorado
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - Beebe Medical Center, Lewes, Delaware
  - Christiana Gynecologic Oncology LLC, Newark, Delaware
  - Delaware Clinical and Laboratory Physicians PA, Newark, Delaware
  - Helen F. Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Regional Hematology and Oncology PA, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - Nanticoke Memorial Hospital, Seaford, Delaware
  - Christiana Care Health System-Wilmington Hospital, Wilmington, Delaware
  - Morton Plant Hospital, Clearwater, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Oncare Hawaii Inc-POB II, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Kuakini Medical Center, Honolulu, Hawaii
  - OnCare Hawaii, Incorporated-Kuakini, Honolulu, Hawaii
  - OnCare Hawaii-Liliha, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Liliha, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Wilcox Memorial Hospital and Kauai Medical Clinic, Lihue, Hawaii
  - Oncare Hawaii, Incorporated-Pali Momi, ‘Aiea, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - The Cancer Center of Hawaii-Leeward, ‘Ewa Beach, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Kootenai Medical Center, Coeur d'Alene, Idaho
  - Kootenai Cancer Center, Post Falls, Idaho
  - Kootenai Cancer Clinic, Sandpoint, Idaho
  - Saint Joseph Medical Center, Bloomington, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Memorial Hospital of Carbondale, Carbondale, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - University of Illinois, Chicago, Illinois
  - Cancer Care Specialists of Central Illinois, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Radiation Oncology of Northern Illinois, Ottawa, Illinois
  - OSF Saint Francis Radiation Oncology at Pekin Cancer Treatment Center, Pekin, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - OSF Saint Francis Radiation Oncology at Peoria Cancer Center, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Central Illinois Hematology Oncology Center, Springfield, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Cancer Care Specialists of Illinois-Swansea, Swansea, Illinois
  - IU Health West Hospital, Avon, Indiana
  - IU Health North Hospital, Carmel, Indiana
  - IU Health Central Indiana Cancer Centers-Fishers, Fishers, Indiana
  - Indiana University-Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - IU Health Methodist Hospital, Indianapolis, Indiana
  - Sidney and Lois Eskenazi Hospital, Indianapolis, Indiana
  - Memorial Regional Cancer Center-Day Road, Mishawaka, Indiana
  - Saint Joseph Regional Medical Center-Mishawaka, Mishawaka, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Michiana Hematology Oncology PC-South Bend, South Bend, Indiana
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic PC-William R Bliss Cancer Center, Ames, Iowa
  - McFarland Clinic PC-Boone, Boone, Iowa
  - Medical Oncology and Hematology Associates-West Des Moines, Clive, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - Alegent Health Mercy Hospital, Council Bluffs, Iowa
  - Greater Regional Medical Center, Creston, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Iowa-Wide Oncology Research Coalition NCORP, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Des Moines, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Laurel, Des Moines, Iowa
  - Mercy Medical Center-Des Moines, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - McFarland Clinic PC-Trinity Cancer Center, Fort Dodge, Iowa
  - McFarland Clinic PC-Jefferson, Jefferson, Iowa
  - McFarland Clinic PC-Marshalltown, Marshalltown, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - Methodist West Hospital, West Des Moines, Iowa
  - Menorah Medical Center, Overland Park, Kansas
  - Saint Luke's South Hospital, Overland Park, Kansas
  - Kansas City NCI Community Oncology Research Program, Prairie Village, Kansas
  - Flaget Memorial Hospital, Bardstown, Kentucky
  - Commonwealth Cancer Center-Corbin, Corbin, Kentucky
  - Saint Elizabeth Medical Center South, Edgewood, Kentucky
  - Saint Elizabeth-Fort Thomas, Fort Thomas, Kentucky
  - Saint Joseph Radiation Oncology Resource Center, Lexington, Kentucky
  - Saint Joseph Hospital East, Lexington, Kentucky
  - Jewish Hospital, Louisville, Kentucky
  - The James Graham Brown Cancer Center at University of Louisville, Louisville, Kentucky
  - Saints Mary and Elizabeth Hospital, Louisville, Kentucky
  - Jewish Hospital Medical Center Northeast, Louisville, Kentucky
  - Jewish Hospital Medical Center South, Shepherdsville, Kentucky
  - Eastern Maine Medical Center, Bangor, Maine
  - Eastern Maine Medical Center Cancer Care, Brewer, Maine
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Saint Agnes Hospital, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Dana-Farber/Brigham and Women's Cancer Center at South Shore, South Weymouth, Massachusetts
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Saint John Hospital and Medical Center, Detroit, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Mercy Health Saint Mary's, Grand Rapids, Michigan
  - Spectrum Health at Butterworth Campus, Grand Rapids, Michigan
  - Allegiance Health, Jackson, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - Saint Mary Mercy Hospital, Livonia, Michigan
  - Mercy Health Mercy Campus, Muskegon, Michigan
  - Saint Joseph Mercy Oakland, Pontiac, Michigan
  - William Beaumont Hospital-Royal Oak, Royal Oak, Michigan
  - Saint Mary's of Michigan, Saginaw, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - William Beaumont Hospital-Troy, Troy, Michigan
  - Saint John Macomb-Oakland Hospital, Warren, Michigan
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Fairview-Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital-Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - Coborn Cancer Center at Saint Cloud Hospital, Saint Cloud, Minnesota
  - Saint Cloud Hospital, Saint Cloud, Minnesota
  - Metro Minnesota Community Oncology Research Consortium, Saint Louis Park, Minnesota
  - Park Nicollet Clinic-Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology and Hematology PA-Woodbury, Woodbury, Minnesota
  - Parkland Health Center-Bonne Terre, Bonne Terre, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Southeast Cancer Center, Cape Girardeau, Missouri
  - Centerpoint Medical Center LLC, Independence, Missouri
  - Capital Region Medical Center-Goldschmidt Cancer Center, Jefferson City, Missouri
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Heartland Hematology and Oncology Associates Incorporated, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - Saint Luke's East-Lee's Summit, Lee's Summit, Missouri
  - Liberty Radiation Oncology Center, Liberty, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - Missouri Baptist Outpatient Center-Sunset Hills, Sunset Hills, Missouri
  - Montana Cancer Consortium NCORP, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Healthcare-Sletten Cancer Institute, Great Falls, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Community Medical Hospital, Missoula, Montana
  - Saint Patrick Hospital-Community Hospital, Missoula, Montana
  - CHI Health Saint Francis, Grand Island, Nebraska
  - Heartland Hematology and Oncology, Kearney, Nebraska
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Saint Elizabeth Regional Medical Center, Lincoln, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Hematology and Oncology Consultants PC, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Alegent Health Lakeside Hospital, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - Midlands Community Hospital, Papillion, Nebraska
  - Cancer and Blood Specialists-Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Henderson, Henderson, Nevada
  - Las Vegas Cancer Center-Henderson, Henderson, Nevada
  - 21st Century Oncology-Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Southeast Henderson, Henderson, Nevada
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Cancer and Blood Specialists-Shadow, Las Vegas, Nevada
  - Nevada Cancer Research Foundation NCORP, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Central, Las Vegas, Nevada
  - 21st Century Oncology-Fort Apache, Las Vegas, Nevada
  - 21st Century Oncology, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Maryland Parkway, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-San Martin, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Southeast, Las Vegas, Nevada
  - Cancer Therapy and Integrative Medicine, Las Vegas, Nevada
  - 21st Century Oncology-Vegas Tenaya, Las Vegas, Nevada
  - Cancer and Blood Specialists-Tenaya, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada-Northwest, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Tenaya, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada-Summerlin, Las Vegas, Nevada
  - Cancer and Blood Specialists-Fort Apache, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Las Vegas Cancer Center-Medical Center, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Centennial Hills, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada-Central Valley, Las Vegas, Nevada
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Memorial Sloan Kettering Cancer Center-Basking Ridge, Basking Ridge, New Jersey
  - Saint Peter's University Hospital, New Brunswick, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Lovelace Women's Hospital, Albuquerque, New Mexico
  - Memorial Sloan Kettering Cancer Center-Commack, Commack, New York
  - Memorial Sloan Kettering Cancer Center-West Harrison, Harrison, New York
  - North Shore University Hospital, Manhasset, New York
  - North Shore-LIJ Health System/Center for Advanced Medicine, New Hyde Park, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Vassar Brothers Medical Center, Poughkeepsie, New York
  - University of Rochester, Rochester, New York
  - Memorial Sloan Kettering Cancer Center-Rockville Centre, Rockville Centre, New York
  - Memorial Sloan Kettering Cancer Center-Sleepy Hollow, Sleepy Hollow, New York
  - Randolph Hospital, Asheboro, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Levine Cancer Institute-Tryon, Charlotte, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Carolina Surgical Clinic of Charlotte PA, Charlotte, North Carolina
  - Oncology Specialists of Charlotte, Charlotte, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute-Pineville, Charlotte, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute-University, Charlotte, North Carolina
  - Southern Oncology Specialists-Charlotte, Charlotte, North Carolina
  - Levine Cancer Institute-Ballantyne, Charlotte, North Carolina
  - CaroMont Breast Surgical Specialists-Gastonia, Gastonia, North Carolina
  - CaroMont Regional Medical Center, Gastonia, North Carolina
  - Cone Health Cancer Center, Greensboro, North Carolina
  - Lake Norman Hematology Oncology Specialists-Huntersville, Huntersville, North Carolina
  - Southern Oncology Specialists-Huntersville, Huntersville, North Carolina
  - Matthews Radiation Oncology Center, Matthews, North Carolina
  - Novant Health Cancer Specialists-Matthews, Matthews, North Carolina
  - Carolinas HealthCare System Union, Monroe, North Carolina
  - Lake Norman Hematology Oncology Specialists-Mooresville, Mooresville, North Carolina
  - Annie Penn Memorial Hospital, Reidsville, North Carolina
  - Strecker Cancer Center-Belpre, Belpre, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - The Christ Hospital, Cincinnati, Ohio
  - Good Samaritan Hospital-Cincinnati, Cincinnati, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio
  - TriHealth Cancer Institute-Westside, Cincinnati, Ohio
  - TriHealth Cancer Institute-Anderson, Cincinnati, Ohio
  - University of Cincinnati, Cincinnati, Ohio
  - Mount Carmel East Hospital, Columbus, Ohio
  - Columbus Oncology and Hematology Associates Inc, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Columbus NCI Community Oncology Research Program, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Delaware Health Center-Grady Cancer Center, Delaware, Ohio
  - Delaware Radiation Oncology, Delaware, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - OhioHealth MedCentral Hospital, Mansfield, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - OhioHealth Marion General Hospital, Marion, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Newark Radiation Oncology, Newark, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - University Pointe, West Chester, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Oregon Health and Science University, Portland, Oregon
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Lehigh Valley Hospital-Muhlenberg, Bethlehem, Pennsylvania
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - Roger Williams Medical Center, Providence, Rhode Island
  - Hilton Head Regional Medical Center, Hilton Head Island, South Carolina
  - Levine Cancer Institute-Rock Hill, Rock Hill, South Carolina
  - Lexington Medical Center, West Columbia, South Carolina
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Memorial Hospital, Chattanooga, Tennessee
  - Pulmonary Medicine Center of Chattanooga-Hixson, Hixson, Tennessee
  - Memorial GYN Plus, Ooltewah, Tennessee
  - Texas Tech University Health Sciences Center-Amarillo, Amarillo, Texas
  - Parkland Memorial Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - M. D. Anderson Cancer Center, Houston, Texas
  - The Methodist Hospital System, Houston, Texas
  - Doctor's Hospital of Laredo, Laredo, Texas
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - Central Vermont Medical Center, Berlin Corners, Vermont
  - University of Vermont College of Medicine, Burlington, Vermont
  - Norris Cotton Cancer Center-North, Saint Johnsbury, Vermont
  - Mary Washington Hospital, Fredericksburg, Virginia
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - Harrison HealthPartners Hematology and Oncology-Bremerton, Bremerton, Washington
  - Harrison Medical Center, Bremerton, Washington
  - Highline Medical Center-Main Campus, Burien, Washington
  - Saint Elizabeth Hospital, Enumclaw, Washington
  - Saint Francis Hospital, Federal Way, Washington
  - Saint Clare Hospital, Lakewood, Washington
  - Harrison HealthPartners Hematology and Oncology-Poulsbo, Poulsbo, Washington
  - Virginia Mason Medical Center, Seattle, Washington
  - Franciscan Research Center-Northwest Medical Plaza, Tacoma, Washington
  - Northwest Medical Specialties PLLC, Tacoma, Washington
  - Green Bay Oncology at Saint Vincent Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital, Green Bay, Wisconsin
  - Green Bay Oncology Limited at Saint Mary's Hospital, Green Bay, Wisconsin
  - Saint Mary's Hospital, Green Bay, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Froedtert and the Medical College of Wisconsin, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Westfields Hospital/Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - Vince Lombardi Cancer Clinic-Oshkosh, Oshkosh, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
  - Big Horn Basin Cancer Center, Cody, Wyoming
  - Billings Clinic-Cody, Cody, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming

REFERENCES:
- [Derived] Boughey JC, Rosenkranz KM, Ballman KV, McCall L, Haffty BG, Cuttino LW, Kubicky CD, Le-Petross HT, Giuliano AE, Van Zee KJ, Hunt KK, Hahn OM, Carey LA, Partridge AH. Local Recurrence After Breast-Conserving Therapy in Patients With Multiple Ipsilateral Breast Cancer: Results From ACOSOG Z11102 (Alliance). J Clin Oncol. 2023 Jun 10;41(17):3184-3193. doi: 10.1200/JCO.22.02553. Epub 2023 Mar 28. PMID 36977292
- [Derived] Cuttino LW, McCall L, Kubicky C, Ballman KV, Le-Petross H, Hunt KK, Haffty B, Rosenkranz KM, Boughey JC. The Feasibility of Radiation Therapy after Breast-Conserving Surgery for Multiple Ipsilateral Breast Cancer: An Initial Report from ACOSOG Z11102 (Alliance) Trial. Int J Radiat Oncol Biol Phys. 2022 Mar 1;112(3):636-642. doi: 10.1016/j.ijrobp.2021.09.054. Epub 2021 Oct 8. PMID 34634438
- [Derived] Rosenkranz KM, Ballman K, McCall L, McCarthy C, Kubicky CD, Cuttino L, Hunt KK, Giuliano A, Van Zee KJ, Haffty B, Boughey JC. Cosmetic Outcomes Following Breast-Conservation Surgery and Radiation for Multiple Ipsilateral Breast Cancer: Data from the Alliance Z11102 Study. Ann Surg Oncol. 2020 Nov;27(12):4650-4661. doi: 10.1245/s10434-020-08893-w. Epub 2020 Jul 22. PMID 32699926
- [Derived] Rosenkranz KM, Ballman K, McCall L, Kubicky C, Cuttino L, Le-Petross H, Hunt KK, Giuliano A, Van Zee KJ, Haffty B, Boughey JC. The Feasibility of Breast-Conserving Surgery for Multiple Ipsilateral Breast Cancer: An Initial Report from ACOSOG Z11102 (Alliance) Trial. Ann Surg Oncol. 2018 Oct;25(10):2858-2866. doi: 10.1245/s10434-018-6583-6. Epub 2018 Jul 9. PMID 29987605

RESULTS

PARTICIPANT FLOW:
Groups:
- Breast Conservation Surgery and Radiation Therapy: Patients undergo breast conserving surgery. Patients receive adjuvant chemotherapy at the physician's discretion. Patients receiving chemotherapy will start treatment within 12 weeks following surgery. Patients receive radiation therapy within 8 weeks following the last dose of chemotherapy or within 10 weeks following surgery if not receiving chemotherapy. Patients receive endocrine therapy at the physician's discretion. Patient observation will occur every 6 months until 5 years after the end of radiation therapy.>> >> therapeutic conventional surgery>>
  >> whole breast irradiation
Period: Overall Study
Arm/Group | Breast Conservation Surgery and Radiation Therapy
Started | 270
Completed | 204
Not Completed | 66
Not completed — Ineligible | 34
Not completed — Converted to mastectomy | 14
Not completed — Unable to achieve negative margins | 2
Not completed — Withdrawal by Subject | 16

BASELINE CHARACTERISTICS:
Arm/Group | Breast Conservation Surgery and Radiation Therapy
Number analyzed (Participants) | 270
Age, Continuous [Median (Full Range); unit: years] | 60.5 [40 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 270
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9
  Not Hispanic or Latino | 245
  Unknown or Not Reported | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 22
  White | 232
  More than one race | 0
  Unknown or Not Reported | 11

OUTCOME MEASURES:

1. Primary Outcome: Local Recurrence
Description: Local recurrence(LR) defined as histologic evidence of ductal carcinoma in situ or invasive breast cancer in the ipsilateral breast or chest wall assessed up to 5 years. The estimated 5-year cumulative incidence of LR will be reported as a percentage of patients expected to experience a LR at 5 years.
Time Frame: 5 years
Population: All patients that received protocol therapy and were evaluated for response
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Breast Conservation Surgery and Radiation Therapy
Number analyzed (Participants) | 204
percentage of participants | 3.1 [1.3 to 6.4]

2. Secondary Outcome: Conversion Rate to Mastectomy
Description: The conversion rate to mastectomy secondary to persistent positive margins; poor cosmesis within the first year of attempting BCS; or inability to satisfy the radiation dose constraints on the boost to the lumpectomy bed of each site of disease.
Time Frame: 5 years
Population: There are only 198 patients in this analysis because it excludes those registered postoperatively
Measure: Number; unit: percentage of patients converted
Groups:
- Breast Conservation Surgery and Radiation Therapy: Patients undergo breast conserving surgery. Patients receive adjuvant chemotherapy at the physician's discretion. Patients receiving chemotherapy will start treatment within 12 weeks following surgery. Patients receive radiation therapy within 8 weeks following the last dose of chemotherapy or within 10 weeks following surgery if not receiving chemotherapy. Patients receive endocrine therapy at the physician's discretion. Patient observation will occur every 6 months until 5 years after the end of radiation therapy.> >>
  >
  >> therapeutic conventional surgery>
  >>
  >
  >> whole breast irradiation
Arm/Group | Breast Conservation Surgery and Radiation Therapy
Number analyzed (Participants) | 198
percentage of patients converted | 7.1

3. Secondary Outcome: Type and Severity of Adverse Effects of Breast-conserving Surgery and Radiation as Assessed by the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0
Time Frame: Up to 30 days post-treatment
Reporting Status: Not Posted

4. Secondary Outcome: Radiation-related Side Effects
Description: Radiation-related side effects of whole-breast radiation with a boost to 1 large or > 1 lumpectomy site as assessed by NCI CTCAE version 4.0.
Time Frame: 17 months
Population: All eligible patients that received radiation therapy.
Measure: Count of Participants; unit: Participants
Arm/Group | Breast Conservation Surgery and Radiation Therapy
Number analyzed (Participants) | 195
Participants
  Grade 1 | 69
  Grade 2 | 74
  Grade 3 | 6

5. Secondary Outcome: Patient's Perception of Cosmesis
Description: Patient's perception of cosmesis will be assessed at their initial post-operative visit as well as 24 months following completion of WBI using the BREAST-Q subscales: satisfaction with breasts, satisfaction with overall outcome, and physical well-being. Patients registered after surgery will not partake in the pre-operative assessment but will be asked to complete subsequent cosmesis surveys. The total score for each of these subscales will be determined using the BREAST-Q scoring module (http://www.mskcc.org/mskcc/shared/Breast-Q/scoreBQ.html). The BREAST-Q has multiple domains, and each domain score is obtained by transforming the raw scale item responses with the Q-Score software program. Each domain results in an independent score from 0 to 100 (higher scores indicate greater satisfaction or quality of life).
Time Frame: 24 months
Measure: Number; unit: percentage of patients
Arm/Group | Breast Conservation Surgery and Radiation Therapy
Number analyzed (Participants) | 216
percentage of patients
  Good or excellent (50-100) | 70.6
  Fair (25-50) | 25.7
  Poor (0-25) | 3.7

ADVERSE EVENTS:
Time Frame: Adverse events were followed for a maximum of 17.1 months and mortality was followed for a maximum of 90.6 months.
Description: All patients that were treated and evaluable for adverse events are included in this adverse events summary. All patients that were registered are included in the mortality summary.
Groups:
- Breast Conservation Surgery and Radiation Therapy: whole breast irradiation
Arm/Group | Breast Conservation Surgery and Radiation Therapy
All-Cause Mortality (participants affected / at risk) | 9/270
Serious Adverse Events (participants affected / at risk) | 8/251
Other Adverse Events (participants affected / at risk) | 169/251
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Breast Conservation Surgery and Radiation Therapy (N=251)
Dermatitis radiation (Injury, poisoning and procedural complications) | 5 (5)
Seroma (Injury, poisoning and procedural complications) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1)
Hematoma (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Breast Conservation Surgery and Radiation Therapy (N=251)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Heart failure (Cardiac disorders) | 1 (1)
Eye disorders - Other, specify (Eye disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1)
Edema trunk (General disorders) | 1 (1)
Fatigue (General disorders) | 20 (20)
Localized edema (General disorders) | 4 (4)
Non-cardiac chest pain (General disorders) | 1 (1)
Pain (General disorders) | 8 (9)
Breast infection (Infections and infestations) | 1 (1)
Lung infection (Infections and infestations) | 1 (1)
Skin infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Wound infection (Infections and infestations) | 9 (11)
Bruising (Injury, poisoning and procedural complications) | 5 (5)
Dermatitis radiation (Injury, poisoning and procedural complications) | 145 (146)
Postoperative hemorrhage (Injury, poisoning and procedural complications) | 3 (3)
Seroma (Injury, poisoning and procedural complications) | 50 (56)
Wound dehiscence (Injury, poisoning and procedural complications) | 2 (2)
Weight loss (Investigations) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 3 (3)
Musculoskeletal, conn tissue - Oth spec (Musculoskeletal and connective tissue disorders) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2)
Paresthesia (Nervous system disorders) | 3 (3)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (2)
Tremor (Nervous system disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Breast pain (Reproductive system and breast disorders) | 13 (13)
Reproductive system and breast -Oth spec (Reproductive system and breast disorders) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 3 (3)
Erythroderma (Skin and subcutaneous tissue disorders) | 1 (1)
Pain of skin (Skin and subcutaneous tissue disorders) | 3 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 6 (6)
Skin and subcut tissue disord - Oth spec (Skin and subcutaneous tissue disorders) | 2 (2)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 8 (8)
Skin induration (Skin and subcutaneous tissue disorders) | 2 (2)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1)
Hematoma (Vascular disorders) | 3 (3)
Hypertension (Vascular disorders) | 5 (5)
Hypotension (Vascular disorders) | 1 (1)
Lymphedema (Vascular disorders) | 15 (15)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-11): https://cdn.clinicaltrials.gov/large-docs/43/NCT01556243/Prot_SAP_000.pdf